CLINICAL TRIAL: NCT01303692
Title: Comparison of Bone Mineral Loss in Prostate Cancer Patients Who is Receiving GnRH Agonist and -Plus Anti-androgen Agent
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-OKR-CAS-2010/1
Record Dates: First submitted 2011-02-23; First posted 2011-02-25 (Estimated); Last update posted 2015-01-14 (Estimated); Status verified 2015-01

CONDITIONS: GnRH Agonist Alone vs. GnRH Agonist Plus Anti-androgen Combination Treated Prostate Cancer Patients
Keywords: bone mineral loss; prostate cancer; GnRH agonist alone vs. GnRH agonist plus anti-androgen combination
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- A: Total of 250 prostate cancer patients receiving GnRH agonist
- B: Total of 250 prostate cancer patients receiving GnRH agonist plus anti-androgen agent

SUMMARY:
Comparison of bone mineral loss in prostate cancer patients who is receiving GnRH agonist and -plus anti-androgen agent

DETAILED DESCRIPTION:
MC MD

ELIGIBILITY:
Inclusion Criteria:

* Korean prostate cancer over 50 years old with pathological confirmation
* Patients receiving GnRH antagonist or GnRH agonist plus anti- androgen combination within 6 months since starting.
* Patients measured bone density level before starting to receive hormone therapies above.

Exclusion Criteria:

* Patients who are treated other anti-osteoporosis drugs and who are treated bisphosphate due to BMD T score below -3.0.
* Patients who are hard to be analysed by attach to other bone disease.
* Patients who are hard to be analysed by limitation of chart record according to investigators'discretion.

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Prostate cancer patients who is receiving GnRH agonist and -plus anti-androgen agent
Sampling Method: Probability Sample
Enrollment: 312 (Actual)
Dates: Start 2011-04; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
comparison of bone density before and after hormone therapy | 1 year
comparison of bone density between GnRH agonist alone vs. CAB group | 1 year

SECONDARY OUTCOMES:
correlation between osteoporosis risk factors such as age, weight, history of smoke, history of alcohol and bone density value | 1 year
correlation between osteoporosis risk factors such as age, weight, history of smoke, history of alcohol and bone density value before and after hormone therapy | 1 year
1year comparison of FRAX score before and after hormonal therapy | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Joon Woo Bahn, Study Director — AstraZeneca Korea
Locations (2):
- South Korea (2):
  - Research Site, Seongnam-si, Gyeonggi-do
  - Research Site, Seoul

REFERENCES:
- [Derived] Kim SH, Joung JY, Kim S, Rha KH, Kim HG, Kwak C, Lee JY, Jeon SS, Hong SK, Jeong H, Jo MK, You D, Jeong IG, Hong JH, Kim CS. Comparison of bone mineral loss by combined androgen block agonist versus GnRH in patients with prostate cancer: A 12 month-prospective observational study. Sci Rep. 2017 Mar 6;7:39562. doi: 10.1038/srep39562. PMID 28262724